CLINICAL TRIAL: NCT06403124
Title: Outcome of Operative Management of Posterior Wall of Acetabulum Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chittagong Medical College (Other)
Responsible Party: Principal Investigator, Munshi Foyjul Rabby, Medical officer, Chittagong Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 59.27.00.013.19.PG.09.2023/992
Record Dates: First submitted 2024-04-26; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Posterior Wall of Acetabulum Fracture
Keywords: Posterior wall of acetabulum, operative management
MeSH Terms: interventions — Open Fracture Reduction; Fracture Fixation, Internal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with posterior wall of acetabulum fracture (Experimental)
  Interventions: Procedure: Open reduction and internal fixation

INTERVENTIONS:
Procedure: Open reduction and internal fixation — Open reduction and internal fixation by reconstruction plate and screws

SUMMARY:
Background: Historically, acetabular fractures were treated conservatively which leading to long lasting morbidity like severe pain, limitation of movement and osteoarthritis. Now, evidence suggest surgery for all acetabular fractures for better outcome.

Objectives: To evaluate the clinical and functional outcomes of open reduction and internal fixation of posterior wall of acetabulum fractures.

Methods: This prospective clinical trial was conducted at Chittagong Medical College hospital, Chattogram, from January 2022 to February 2024. Sample size was 32 with fractures as per set criteria and was treated surgically. The outcome variables were functional (according to modified Merle D'Aubigne and Postel score) and radiological (according to Matta's grading). Evaluation was done at 6th weeks and at 03rd, 06th, 09th months. Detailed history, clinical examination, investigations, operative details, post-operative outcome and other parameters were documented. Data were collected in data collection form and were analyzed at the end of the study by using SPSS-25. P-value was considered as statistically significant when it was less than 0.05 and confidence interval was set at 95% level.

ELIGIBILITY:
Inclusion Criteria:

* Posterior wall fracture with unstable hip joint
* Posterior wall fracture with posterior column or transverse fracture
* incarcerated osteochondral fragment
* Age more than 18 years and less than 60 years
* injury within 03 weeks.

Exclusion Criteria:

* open fracture
* associated other acetabular fracture

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Functional outcome | 09 months
  Functional outcome by Modified Merle d'Aubigne-Postel Score, Highest score - 18, that means excellent outcome and lowest score - 03, that means poor outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Chittagong Medical College, Chittagong, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes